CLINICAL TRIAL: NCT00670514
Title: A Comparing Study of the Smoking Cessation Program NIX Individual and the Self-Help Program Fimpa Dig Fri
Brief Title: Smoking Cessation in a Dentistry Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Västmanland County Council, Sweden (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Smoking cessation project
Record Dates: First submitted 2008-04-16; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Smoking
Keywords: RCT; tobacco; treatment intensity; dentistry; follow-up; Smoking cessation; Cost effectiveness
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Nix Individual (Active Comparator): High Treatment Intensity
  Interventions: Behavioral: Nix Individual
- 2 Fimpa dig fri (Placebo Comparator): Low Treatment Intensity
  Interventions: Behavioral: Fimpa dig fri

INTERVENTIONS:
Behavioral: Nix Individual — Eight 40-minutes sessions at the local dental clinic during 4 months. Written material and counseling by a dental hygienist with special training in smoking cessation, according to a fixed program. A traditional smoking cessation program with a mixture of behavior therapy, coaching and pharmacological advises. Two questionnaires.
  Arms: 1 Nix Individual
Behavioral: Fimpa dig fri — One 30-minute counseling session at the local dental clinic, focusing on explaining the content of a traditional self-help program ("Fimpa dig fri"). The leaflet contains an 8-week program with instructions and tasks to perform. Two questionnaires.
  Arms: 2 Fimpa dig fri

SUMMARY:
Aim: to assess relative effectiveness of a high and a low intensity intervention for smoking cessation support in a dental clinic setting.

Method: 300 smokers were randomly assigned to support with either low (LTI) or high treatment intensity (HTI).

Main outcome measures were self-reported point-prevalence and continuous abstinence (≥183 days).

ELIGIBILITY:
Inclusion Criteria:

* Adult daily smokers in the county of Västmanland

Exclusion Criteria:

* Reading difficulties
* Not fluent in the Swedish language

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-04

PRIMARY OUTCOMES:
Point prevalence abstinence

SECONDARY OUTCOMES:
Continuous abstinence

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for clinical research, Central Hospital, Västerås, Sweden

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- [Derived] Nohlert E, Ohrvik J, Tegelberg A, Tillgren P, Helgason AR. Long-term follow-up of a high- and a low-intensity smoking cessation intervention in a dental setting--a randomized trial. BMC Public Health. 2013 Jun 19;13:592. doi: 10.1186/1471-2458-13-592. PMID 23777201
- [Derived] Nohlert E, Tegelberg A, Tillgren P, Johansson P, Rosenblad A, Helgason AR. Comparison of a high and a low intensity smoking cessation intervention in a dentistry setting in Sweden: a randomized trial. BMC Public Health. 2009 Apr 30;9:121. doi: 10.1186/1471-2458-9-121. PMID 19405969